CLINICAL TRIAL: NCT04507542
Title: Playing and Singing for the Recovering Brain: Efficacy of Enriched Social-Motivational Musical Interventions in Stroke Rehabilitation
Brief Title: Enriched Music-Supported Therapy to Restore Motor Deficits After Stroke
Acronym: HOMEMUSIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Barcelona (Other)
Collaborators: Artificial Intelligence Research Institute, Spanish National Research Council (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Antoni Rodriguez Fornells, Research Professor in Catalan Institution for Research and Advanced Studies, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201729.30
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; music therapy
MeSH Terms: conditions — Stroke | interventions — Hand Strength

STUDY DESIGN:
Intervention Model Description: A parallel-group randomised controlled trial will be conducted with participants being randomised to either an enriched Music-Supported Therapy group or to a control treatment group receiving the Graded Repetitive Arm Supplementary Program (GRASP, Harris et al., 2009).
Who Masked: Outcomes Assessor
Masking Description: A clinical researcher with expertise in stroke rehabilitation will perform the evaluations and will be blinded to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched Music-Supported Therapy group (Experimental): Participants in the eMST-group will follow a 10-week program of Enriched Music-Supported Therapy. The program comprises 3 individual self-training sessions and 1 group session per week (total program duration: 40 hours).
  Interventions: Behavioral: Enriched Music-Supported Therapy
- Control group (Active Comparator): Participants in the control intervention group will follow the Graded Repetitive Arm Supplementary Program (GRASP, Harris et al., 2009). They will be asked to complete 4 weekly one-hour session for 10 weeks (total program duration: 40 hours).
  Interventions: Behavioral: Graded Repetitive Arm Supplementary Program

INTERVENTIONS:
Behavioral: Enriched Music-Supported Therapy — Home-based rehabilitation program for stroke patients aimed at improving the upper extremity motor function. The program is based on musical training, combining self-training sessions of music playing using an app for electronic tablets and music therapy group sessions.
  Other Names: Music-Supported Therapy
  Arms: Enriched Music-Supported Therapy group
Behavioral: Graded Repetitive Arm Supplementary Program — Home-based rehabilitation program for stroke patients aimed at improving the upper extremity motor function. The program comprises self-training sessions of mass repetition of movements and task-specific exercises for the upper extremity.
  Other Names: GRASP
  Arms: Control group

SUMMARY:
Music-Supported Therapy (MST) is a rehabilitation technique to improve the upper extremity motor function of stroke patients through playing musical instruments. A modified version of the MST protocol has been created (hereafter, referred as enriched MST, eMST) to include (i) a home-based self-training program using an app for electronic tablets and (ii) weekly group sessions of musical playing strengthening the motivational and emotional components of music playing. A randomised controlled trial will be conducted to test the effectiveness of this enriched MST (eMST) protocol in improving motor functions, cognition, emotional well-being and quality of life when compared to a program of home-based exercises utilizing the Graded Repetitive Arm Supplementary Program (GRASP). Sixty stroke patients will be recruited and randomly allocated to an eMST group (n=30) or a control GRASP intervention group (n=30). Patients will be evaluated before and after a 10-week intervention, as well as at 3-month follow-up. The primary outcome of the study is the functionality of the paretic upper limb measured with the Action Research Arm Test. Secondary outcomes include other motor and cognitive functions, emotional well-being and quality of life measures as well as self-regulation and self-efficacy outcomes. We hypothesize that patients treated with eMST will show larger improvements in their motor and cognitive functions, emotional well-being and quality of life than patients treated with a home-based GRASP intervention.

ELIGIBILITY:
Inclusion criteria:

* Presence of mild-to-moderate paresis of the upper extremity after a stroke (having a score between 1 and 4 in the Medical Research Council Scale for Muscle Strength at the distal muscles of the upper extremity);
* More than 6 months post-stroke;
* Completion of formal rehabilitation programs.

Exclusion criteria:

* Major language or cognitive deficits affecting comprehension (Mini-Mental State Examination < 24);
* Neurological or psychiatric co-morbidity;
* Other musculoskeletal condition affecting upper extremity motor function (e.g. fracture or arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Action Research Arm Test | immediately after the intervention
  Upper extremity function measure. The measure is a 19-item test divided into four subtests (grasp, grip, pinch and gross movement). For each item, the patient is asked to perform a simple task that involves a functional movement of the affected upper limb. Each task is rated using a 4-point ordinal scale. The maximum possible score is 57 and the minimal clinically important difference is 5.7 points.
Change in Action Research Arm Test | 3 months after completing the intervention
  Upper extremity function measure. The measure is a 19-item test divided into four subtests (grasp, grip, pinch and gross movement). For each item, the patient is asked to perform a simple task that involves a functional movement of the affected upper limb. Each task is rated using a 4-point ordinal scale. The maximum possible score is 57 and the minimal clinically important difference is 5.7 points.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment of Motor Recovery after Stroke | immediately after the intervention
  Motor impairment measure. It comprises 33 items that evaluate motor impairment in the affected upper limb. The test is divided into 4 sections (shoulder, forearm and elbow, wrist, hand and coordination) assessing reflexes, flexor and extensor synergies, range of motion, and overall coordination and speed of the upper extremity. Each item is graded using an ordinal scale from 0 to 2. The maximum possible score is 66 and the minimal clinically important difference for chronic stroke patients is 5.2 points.
Change in Fugl-Meyer Assessment of Motor Recovery after Stroke | 3 months after completing the intervention
  Motor impairment measure. It comprises 33 items that evaluate motor impairment in the affected upper limb. The test is divided into 4 sections (shoulder, forearm and elbow, wrist, hand and coordination) assessing reflexes, flexor and extensor synergies, range of motion, and overall coordination and speed of the upper extremity. Each item is graded using an ordinal scale from 0 to 2. The maximum possible score is 66 and the minimal clinically important difference for chronic stroke patients is 5.2 points.
Change in Grip Strength in Kgs | immediately after the intervention
  Grip strength measure, Biometrics E-Link tool
Change in Grip Strength in Kgs | 3 months after completing the intervention
  Grip strength measure, Biometrics E-Link tool
Change in Box and Block Test | immediately after the intervention
  Gross manual dexterity measure
Change in Box and Block Test | 3 months after completing the intervention
  Gross manual dexterity measure
Change in Nine Hole Pegboard Test | immediately after the intervention
  Fine manual dexterity measure
Change in Nine Hole Pegboard Test | 3 months after completing the intervention
  Fine manual dexterity measure
Change in Chedoke Arm and Hand Activity Inventory | immediately after the intervention
  Motor performance in activities of daily living measure. The test is composed of 13 different tasks (i.e. open a jar of coffee, make a phone call, clean a pair of eyeglasses) and each task is graded using an ordinal scale from 1 to 7. Maximum score is 91, indicating good performance.
Change in Chedoke Arm and Hand Activity Inventory | 3 months after completing the intervention
  Motor performance in activities of daily living measure. The test is composed of 13 different tasks (i.e. open a jar of coffee, make a phone call, clean a pair of eyeglasses) and each task is graded using an ordinal scale from 1 to 7. Maximum score is 91, indicating good performance.
Change in Behaviour Rating Inventory of Executive Function | immediately after the intervention
  Executive function measure. It comprises 75 items describing various behaviours, and the participant is asked to report if the behaviour is never a problem, sometimes a problem or often a problem.
Change in Behaviour Rating Inventory of Executive Function | 3 months after completing the intervention
  Executive function measure. It comprises 75 items describing various behaviours, and the participant is asked to report if the behaviour is never a problem, sometimes a problem or often a problem.
Change in Sustained Attention to Response Task | immediately after the intervention
  Sustained attention measure
Change in Sustained Attention to Response Task | 3 months after completing the intervention
  Sustained attention measure
Change in Figural Memory Subtest | immediately after the intervention
  Visuospatial memory measure
Change in Figural Memory Subtest | 3 months after completing the intervention
  Visuospatial memory measure
Change in Rey Auditory Verbal Learning Test | immediately after the intervention
  Verbal learning measure
Change in Rey Auditory Verbal Learning Test | 3 months after completing the intervention
  Verbal learning measure
Change in Fluency Test | immediately after the intervention
  Verbal fluency measure
Change in Fluency Test | 3 months after completing the intervention
  Verbal fluency measure
Change in Beck Depression Inventory-II | immediately after the intervention
  Depression measure. It comprises 21 multiple-choice questions that are scored on a scale from 0 to 3. The participant is asked about feelings, thoughts and behaviours of the past week. Higher scores indicate depression severity and the maximum possible score of the measure is 63.
Change in Beck Depression Inventory-II | 3 months after completing the intervention
  Depression measure. It comprises 21 multiple-choice questions that are scored on a scale from 0 to 3. The participant is asked about feelings, thoughts and behaviours of the past week. Higher scores indicate depression severity and the maximum possible score of the measure is 63.
Change in Apathy Evaluation Scale | immediately after the intervention
  Apathy measure. The scale comprises a self and informant reports both consisting of 18 items that are scored on a 4-point Likert scale, where higher scores indicate more apathy.
Change in Apathy Evaluation Scale | 3 months after completing the intervention
  Apathy measure. The scale comprises a self and informant reports both consisting of 18 items that are scored on a 4-point Likert scale, where higher scores indicate more apathy.
Change in Profile of Mood States | immediately after the intervention
  Mood measure. The measure includes 65 items that are scored on a 5-point Likert scale ranging from 0 "not at all" to 4 "extremely".
Change in Profile of Mood States | 3 months after completing the intervention
  Mood measure. The measure includes 65 items that are scored on a 5-point Likert scale ranging from 0 "not at all" to 4 "extremely".
Change in Stroke Impact Scale | immediately after the intervention
  Quality of life measure. It is a 59-item self-report questionnaire that assesses muscle strength, hand function, basic and instrumental activities of daily living, global mobility, communication, emotion, memory and thinking, and participation.
Change in Stroke Impact Scale | 3 months after completing the intervention
  Quality of life measure. It is a 59-item self-report questionnaire that assesses muscle strength, hand function, basic and instrumental activities of daily living, global mobility, communication, emotion, memory and thinking, and participation.

OTHER OUTCOMES:
Treatment Self-regulation Questionnaire | Baseline
  Self-regulation measure. It evaluates the type of self-regulation (external, interjected, identified or intrinsic) or motivation (external or intrinsic) of the participants to engage with the rehabilitation program. It is a 15-item self-report questionnaire scored on a 7-point scale (1: not all true; 4: somewhat true; 7: very true).
Treatment Questionnaire Concerning Continued Program | Week 5 (after the first half of the intervention)
  Self-regulation measure. It is a 15-item self-report questionnaire scored on a 7-point scale (1: not all true; 4: somewhat true; 7: very true).
Intrinsic Motivation Inventory | immediately after the intervention
  Motivation measure. It consists of 24 self-report questions divided into six different psychological constructs reflecting positive or negative predictors of intrinsic motivation: 1) interest/enjoyment; 2) perceived competence; 3) effort/importance; 4) pressure/tension; 5) perceived choice; and 6) value/usefulness. It is scored on a 7-point scale (1: not all true; 4: somewhat true; 7: very true).
Strategies Used to Promote Health Questionnaire | Baseline
  Self-efficacy measure. It is a 29-item self-report questionnaire that evaluates the degree of self-care and self-efficacy through four factors consistent with the underlying self-efficacy theory upon which the scale is based: 1) coping, 2) stress reduction, 3) making decisions, and 4) enjoying life. It is scored on a 5-point scale (from 1: very little confidence to 5: quite a lot of confidence).

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Rodríguez Fornells, PhD, Principal Investigator — Bellvitge Biomedical Research Institute, University of Barcelona; Jennifer Grau Sánchez, PhD, Study Director — Bellvitge Biomedical Research Institute, University of Barcelona
Locations (1):
- Bellvitge Biomedical Research Institute, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Segura E, Grau-Sanchez J, Cerda-Company X, Porto MF, De la Cruz-Puebla M, Sanchez-Pinsach D, Cerquides J, Duarte E, Palumbo A, Turry A, Raghavan P, Sarkamo T, Munte TF, Arcos JL, Rodriguez-Fornells A. Enriched music-supported therapy for individuals with chronic stroke: a randomized controlled trial. J Neurol. 2024 Oct;271(10):6606-6617. doi: 10.1007/s00415-024-12570-3. Epub 2024 Aug 7. PMID 39112892
- [Derived] Grau-Sanchez J, Segura E, Sanchez-Pinsach D, Raghavan P, Munte TF, Palumbo AM, Turry A, Duarte E, Sarkamo T, Cerquides J, Arcos JL, Rodriguez-Fornells A. Enriched Music-supported Therapy for chronic stroke patients: a study protocol of a randomised controlled trial. BMC Neurol. 2021 Jan 12;21(1):19. doi: 10.1186/s12883-020-02019-1. PMID 33435919
- See also: Research group webpage — http://www.brainvitge.org